CLINICAL TRIAL: NCT03540056
Title: Testicular Growth During Puberty in Boys With and Without a Left-sided Varicocele
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Donald Vaganée, Principal Investigator, Universiteit Antwerpen
Other Study IDs: B300201730926
Record Dates: First submitted 2018-05-03; First posted 2018-05-30 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Varicocele; Scrotal Disorder
Keywords: varicocele; testicular growth
MeSH Terms: conditions — Varicocele | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Boys without varicocele: Boys thoroughly examined but without diagnose of varicocele
  Interventions: Diagnostic Test: Ultrasound
- Boys with a varicocoele: Boys with a diagnosed varicocele of any stage possible.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — We use ultrasound to measure the PRF and the testicular volumes.

SUMMARY:
Prospective observational study.

A varicocele is defined as a dilatation of the veins in the plexus pampiniformis in the testicles. Varicoceles are a diagnostic dilemma and a therapeutic challenge. Most of the boys with a varicocele don't show any symptoms, but approximately 15-20% experience some sort of infertility later during their life. There still isn't any consensus on when treating the patient is the right choice. Reliable scientific research about parameters able to predict the later stages of the boy with a varicocele is therefore needed. The purpose of this study is to how testicular growth could predict the outcome of boys with a varicocele.

During this study, testicular growth in boys with and without a left-sided varicocele will be examined in different schools using ultrasound to measure the testicular volumes, the PRF and the TAI to be able to collect sufficient data with the purpose to be able to predict whether testicular growth is a significant predictor on the progression of a varicocele.

ELIGIBILITY:
Inclusion Criteria:

1. Boys aged 11-16 years without any evidence of a current or past pathology influencing testicular growth

Exclusion Criteria:

1. Boys with a current or past inguinoscrotal pathology (varicocele, testicular microlithiasis, cryptorchidism, retractile testis, orchidectomy, testicular torsion, orchitis or epididymitis, hypospadias, inguinal hernia, oeprated varicocele, hydrocele and epididymal cysts)
2. Boys with evidence of disorders influencing testicular growth (e.g. growth disorders)
3. Boys with missing or incomplete data on Tanner stages for genital development
4. Boys with a psychiatric disorder

Ages: 11 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: The study population consists of adolescent boys with or without a varicocele being between the age 11 and 16 years old when enlisting in the study. Recruitment took place at the Antwerp University Hospital and through medical checkups in secondary schools in Antwerp and West-Flanders.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2012-10-10 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Change in testicular volumes in adolescents boys | 3 years
  Scrotal ultrasound is performed to assess testicular dimensions after which testicular volume is calculated. Multiple measurements are performed over a time period of 3 years.
Chang in haemodynamic parameters in adolescent boys with a varicocele | 3 years
  Scrotal doppler ultrasound is performed and the peak retrograde flow is determined. Multiple measurements are performed over a time period of 3 years.

SECONDARY OUTCOMES:
Semen analysis in varicoele patients | After liquefaction (30-35 minutes after ejaculation)
  Routine standard semen analysis as well as DNA fragmentation testing.

CONTACTS AND LOCATIONS:
Overall Officials: Gunter De Win, MD PhD FEABU, Study Director — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No